CLINICAL TRIAL: NCT06904027
Title: A Single-arm, Prospective, Multi-center Post-market Clinical Study of Glycerol Phenylbutyrate in Chinese Patients With Urea Cycle Disorders
Brief Title: A Clinical Study of Glycerol Phenylbutyrate in Chinese Patients With Urea Cycle Disorders
Status: Recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Xiaoping Luo, Professor, Tongji Hospital
Other Study IDs: WH002A401
Record Dates: First submitted 2025-03-10; First posted 2025-04-01 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Urea Cycle Disorders
Keywords: Chinese; Pediatric patients; Urea cycle disorders; Glycerol phenylbutyrate
MeSH Terms: conditions — Urea Cycle Disorders, Inborn | interventions — glycerol phenylbutyrate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Glycerol phenylbutyrate cohort: Glycerol Phenylbutyrate was used.
  Interventions: Drug: Glycerol phenylbutyrate Oral Liquid

INTERVENTIONS:
Drug: Glycerol phenylbutyrate Oral Liquid — Administration and dosage: The recommended total daily dose of glycerol phenylbutyrate is calculated based on the patient's body surface area, ranging from 4.5 mL/m2/d to 11.2 mL/m2/d:
  1. Recommended initial dose in phenylbutyrate-naïve patients
     * Patients with body surface area (BSA) < 1.3 m2: 8.5 mL/m2/day
     * Patients with body surface area (BSA) ≥ 1.3 m2: 7 mL/m2/day
  2. Initial dose for patients switching from sodium phenylbutyrate to glycerol phenylbutyrate: Total daily dose of glycerol phenylbutyrate (ml) = total daily dose of sodium phenylbutyrate granules (g) ×0.81 Medication Schedule: The daily total dose should be divided into equal amounts and administered with each meal or feeding (such as three to six times daily).
  Other Names: HPN-100; GT4P; Glyceryl tri-(4-phenylbutyrate); RAVICTI

SUMMARY:
Urea cycle disorders (UCD) are rare diseases in China, would lead to high mortality and disability, which require long-term management due to the recurrent symptoms. This multi-center, prospective, single-arm study was designed to assess the efficacy and safety of Glycerol Phenylbutyrate for Chinese pediatric patients with UCD, to provide the additional references and treatment options for Chinese UCD patients, and enhance the clinical management of UCD in China. This study primarily observes patients with UCD who are on long-term treatment with glyceryl phenylbutyrate, the total planned observation period is 5 years.

DETAILED DESCRIPTION:
The duration of treatment with GPB in this study was 5 years. Forty participants aged 0-18 years with a diagnosis of UCD, including carbamoyl phosphate synthetase I deficiency, ornithine carbamoyltransferase deficiency, citrullinemia type I, argininosuccinic aciduria, argininemia, or hyperornithinemia-hyperammonemia-homocitrullinuria (HHH) syndrome, and who plan to use and have not used glycerol phenylbutyrate in the previous 3 months (including 3 months) were enrolled. Participants should return to clinic visits at 1 month and 3 months after enrollment. They were queried about any adverse events (AEs), dosage change of the study drug or hyperammonemic crises (HACs) that occurred since the last visit, and blood samples were collected for the analysis of ammonia and blood biochemistry. Then the detailed information on AEs, dosage change of the study drug, HACs, and data about ammonia, routine clinical laboratory safety tests and neurocognitive outcomes that have been actually completed in the clinical practice of the patients will be collected every 6 months until 5 years. Height, weight and/or head circumference data were also collected at each visit. The assessments would be conducted at 1, 3, and 6 months, and subsequently on a semi-annual basis. The evaluation of ammonia levels, frequency of HACs, dosage of the study drug, AEs, serious AEs, and concomitant medications were included. The neurocognitive outcomes, growth and development of the participants would be described at the end.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 0-18 years;
2. Subject and/or subject's legally authorized representative willing to follow the therapeutic regimen, dietary management and visit plan of the study, and voluntarily signing informed consent form;
3. Patients with the following subtypes of UCD: Carbamoyl phosphate synthetase I deficiency, Ornithine translocase deficiency, citrullinemia type I, argininosuccinic aciduria, argininemia, and hyperornithinemia-hyperammonemia-homocitrullinuria (HHH) syndrome;
4. Patients planned to use glycerol phenylbutyrate who have not used it in past 3 months (including at the time of 3 months);
5. Men with fertility and women of childbearing potential (with menstruation) who are willing to take effective contraceptive measures during the period from the date of signing the informed consent to 1 months after the last dose of the study drug, such as abstinence, condoms, intra-uterine contraceptive devices, and double barrier methods (such as condoms + contraceptive diaphragms). Pregnancy test results must be negative for women of childbearing age within ≤ 7 days before the initial administration of study drug.

Exclusion Criteria:

1. Hypersensitivity to any of the active ingredient, including phenylbutyrate (PBA), phenylacetate acid (PAA) and phenylacetyl glutamine (PAGN), or excipients;
2. Use of any drug known to significantly affect renal clearance (such as probenecid) or increase protein catabolism (such as corticosteroids) or other drugs known to increase blood ammonia levels (such as valproate) within 24 h before the first administration;
3. Use of other nitrogen-scavenging agent at the same time after enrollment, such as sodium phenylbutyrate and sodium benzoate;
4. Pregnant or breastfeeding females.
5. Other reasons, in the opinion of the investigator, that may affect the patient's compliance and safety in participating in the study.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Long term treatment for pediatric patients with UCD, aged 0-18 years, who cannot be managed with protein restriction and/or amino acid supplementation alone, including carbamoyl phosphate synthetase I deficiency, ornithine carbamoyltransferase deficiency, citrullinemia type I, argininosuccinic aciduria, argininemia, and hyperornithinemia-hyperammonemia-homocitrullinuria (HHH) syndrome.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Mean blood ammonia levels at month 3 after enrollment. | months 3
  The average of blood ammonia levels at months 3 after enrollment.

SECONDARY OUTCOMES:
Mean blood ammonia levels | Baseline, Month 1, Month 6, and every 6 months thereafter (1-5 years)
  The average of blood ammonia levels at period of baseline, month 1, month 6, and every 6 months thereafter (1-5 years)
Maximum blood ammonia levels | Baseline, Month 1, Month 3, Month 6, and every 6 months thereafter (1-5 years)
  The maximum blood ammonia levels at period of baseline, month 1, month 3, month 6, and every 6 months thereafter (1-5 years)
Frequency of hyperammonaemic crisis | Baseline, Month 1, Month 3, Month 6, and every 6 months thereafter (1-5 years)
  The frequency of hyperammonaemic crisis at period of baseline, month 1, month 3, month 6, and every 6 months thereafter (1-5 years)
Height | Baseline, Month 1, Month 3, Month 6, and every 6 months thereafter (1-5 years).
  The change of height to the baseline in children aged 0-18 years old, and the proportion of weight in the upper, upper-middle, middle, lower-middle, and lower categories for each age group, according to the growth standards for children under 7 years old (WS/T 423-2022) and standard for height level classification among children and adolescents aged 7~18 years (WS/T 612-2018）issued by the National Health Commission of the People's Republic of China.
Weight | Baseline, Month 1, Month 3, Month 6, and every 6 months thereafter (1-5 years)
  The change of weight to the baseline in children aged 0-7 years old, and the proportion of weight in the upper, upper-middle, middle, lower-middle, and lower categories for each age group, according to the growth standards for children under 7 years old issued by the National Health Commission of the People's Republic of China (WS/T 423-2022).
Head circumference | Baseline, Month 1, Month 3, Month 6, and every 6 months thereafter (1-5 years)
  The change of head circumference to the baseline in children aged 0-3 years old, and the proportion of head circumference in the upper, upper-middle, middle, lower-middle, and lower categories for each age group, according to the growth standards for children under 7 years old issued by the National Health Commission of the People's Republic of China (WS/T 423-2022).
Dose adjustment changes | Baseline, Month 1, Month 3, Month 6, and every 6 months thereafter (1-5 years)
  The changes of dose adjustment in glycerol phenylbutyrate throughout the study
Mean Neonatal Behavioral Neurological Assessment Scores: Behavioral ability, passive muscle tone, active muscle tone, primitive reflexes, and general assessment | Month 6, every year thereafter (1-5 years)
  The neonatal behavioral neurological assessment (NBNA) scale was used for newborn participants who were at least 2 months of age, consisting of 20 items, with a maximum score of 40 points. The total scores of the NBNA are derived from the cumulative sum of the scores obtained in behavioral ability (6 items), passive muscle tone (4 items), active muscle tone (4 items), primitive reflexes (3 items), and general assessment (3 items), which are collected according to the scales have been actually completed by the subjects in the clinical practice. The total scores greater than 37 is considered normal, while a score less than or equal to 37 is considered abnormal.
Mean Bayley Scale of Infant Development Scores: mental scale, motor scale | Month 6, every year thereafter (1-5 years)
  The Bayley Scale of Infant Development was used for infant participants whose ages range from 2 months to 30 months, consisting of 244 behavioral items, including 163 items on the mental scale and 81 items on the motor scale. The scores of each infant on the mental and motor scales are converted into standard scores with a mean of 100 and a standard deviation of 16 according to age groups, thereby calculating the Mental Development Index (MDI) and the Psychomotor Development Index (PDI). A total score of MDI and PDI, which are collected according to the scales have been actually completed by the subjects in the clinical practice, are less than 70 indicates developmental delay, 70-79 indicates a borderline state, 80-89 indicates low average, 90-109 indicates average, 110-119 indicates high average, 120-129 indicates superior, and a score of 130 or above indicates very superior.
Mean Gesell Developmental Diagnosis Scale Scores | Month 6, every year thereafter (1-5 years)
  The assessment for Gesell Developmental Diagnosis Scale Scores was used for participants whose ages range from 30 months to 6 years, including five areas: gross motor skills, fine motor skills, adaptive behavior, language, and personal-social behavior. The observed behavioral patterns are identified based on the standard of normal behavioral patterns and are expressed in terms of age. This age is then compared with the actual age to calculate the Developmental Quotient (DQ), which is DQ = Developmental Age / Actual Age × 100, and the values of DQ are collected according to the scales have been actually completed by the subjects in the clinical practice. A DQ of 85 or above is considered normal for the nervous system, a DQ between 75 and 85 (inclusive of 75 but exclusive of 85) indicates a borderline level of nervous system impairment, and a DQ below 75 indicates nervous system damage.
Mean Wechsler Preschool and Primary Scale of Intelligence Scores: The Verbal Intelligence Quotient, the Performance Intelligence Quotient | Month 6, every year thereafter (1-5 years)
  The Chinese - Wechsler Preschool and Primary Scale of Intelligence (C - WYCSI) was used for children participants whose ages range from 4 to 6 years. The Verbal Intelligence Quotient (VIQ) test includes five subtests: Information, Picture Vocabulary, Arithmetic, Picture Comprehension, and Comprehension. The Performance Intelligence Quotient (PIQ) test includes five subtests: Animal Hatching, Picture Completion, Mazes, Geometric Shapes, and Block Design. The intelligence quotient (IQ) score obtained from the 10 subtests of VIQ and PIQ is the Full Intelligence Quotient (FIQ). The values for VIQ, PIQ and FIQ are collected according to the scales have been actually completed by the subjects in the clinical practice. FIQ is divided into five levels: ≥130 is superior, 116 - 129 is above average, 85 - 115 is average, 70 - 84 is below average, and < 70 is intellectual disability.
Mean Wechsler Intelligence Scale for Children Scores: The Verbal Intelligence Quotient, the Performance Intelligence Quotient | Month 6, every year thereafter (1-5 years)
  The Chinese-Wechsler intelligence scale of children (C-WISC）was used for participants whose ages range from 7 to 18 years. This scale consists of 11 subtests. The Verbal Intelligence Quotient (VIQ) test includes Information, Comprehension, Similarities, Arithmetic, Digit Span, and Vocabulary. The Performance Intelligence Quotient (PIQ) test includes Picture Completion, Picture Arrangement, Block Design, Object Assembly, and Coding. First, the raw score is calculated based on the test results of the examinee. Then, the corresponding age-specific scale score coefficient is checked and converted into a scale score. The sum of the VIQ and PIQ scale scores is the full intelligence quotient (FIQ) score, which are collected according to the scales have been actually completed by the subjects in the clinical practice. A FIQ of ≥120 is classified as high intelligence, 90-119 is classified as normal intelligence, and a score < 90 is classified as low intelligence.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Luo, M.D., Principal Investigator — Tongji Hospital
Locations (5):
- China (5):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - Tongji Hosipital, Wuhan, Hubei
  - Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No